CLINICAL TRIAL: NCT06178354
Title: A Pragmatic Phase 2 Study of Focal Ablation (Focal Cryotherapy or High Intensity Frequency Ultrasound) in Men With Clinically Localized Prostate Cancer
Brief Title: Focal Ablation With Focal Cryotherapy or HIFU for the Treatment of Men With Localized Prostate Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Marc Dall'Era, MD (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Marc Dall'Era, MD, Principal Investigator, University of California, Davis
Organization: University of California, Davis (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCDCC306; NCI-2023-09811 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); UCDCC306 (Other: University of California Davis Comprehensive Cancer Center); P30CA093373 (NIH)
Record Dates: First submitted 2023-12-09; First posted 2023-12-21 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Localized Prostate Carcinoma; Stage I Prostate Cancer AJCC v8; Stage II Prostate Cancer AJCC v8; Stage IIIA Prostate Cancer AJCC v8; Stage IIIB Prostate Cancer AJCC v8
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Cryosurgery; High-Intensity Focused Ultrasound Ablation; Extracorporeal Shockwave Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (cryosurgery, high intensity focused ultrasound) (Experimental): Patients undergo focal cryotherapy or high intensity focused ultrasound on study.
  Interventions: Procedure: Cryosurgery; Procedure: High-Intensity Focused Ultrasound Ablation; Other: Survey Administration

INTERVENTIONS:
Procedure: Cryosurgery — Undergo focal cryotherapy ablation
  Other Names: Ablation, Cryo; Cryoablation; cryosurgical ablation
Procedure: High-Intensity Focused Ultrasound Ablation — Undergo high intensity frequency ultrasound ablation
  Other Names: Echopulse; Echotherapy; HIFU; High Intensity Focused Ultrasound; High Intensity Focused Ultrasound Therapy; High-intensity Focused Ultrasound; High-intensity Focused Ultrasound Therapy
Other: Survey Administration — Ancillary studies

SUMMARY:
This clinical trial evaluates the effectiveness of focal ablation with either focal cryotherapy or high intensity frequency ultrasound for the treatment of men with localized prostate cancer. Focal cryotherapy kills tumor cells by freezing them. High intensity frequency ultrasound uses highly focused ultrasound waves to produce heat and destroy tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the efficacy of focal therapy for treatment of prostate cancer.

SECONDARY OBJECTIVES:

I. Patient reported urinary, sexual function and quality of life (QOL) at 1 year.

II. To assess safety.

OUTLINE:

Patients undergo focal cryotherapy or high intensity focused ultrasound on study.

After completion of study treatment, patients are followed up at 7-14 days and periodically for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and willingness to sign an informed consent form
* Clinically localized grade group 1, 2, or 3 prostate cancer and unilateral magnetic resonance imaging (MRI) visible lesion(s). Up to 3 lesions will be allowed for focal treatment
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1 (Karnofsky ≥ 70%)
* Patients ≥ 18 years of age at time of consent
* Life expectancy ≥ 5 years
* Ability and stated willingness to adhere to the study visit schedule and other protocol procedures/requirements for the duration of the study

Exclusion Criteria:

* Nodal or distant metastases
* Prior treatment for prostate cancer
* Anticipated treatment with any cancer intervention, including radiation, hormonal therapy or surgery ≤ 6 months prior to focal therapy in this study
* Known contraindications to general anesthesia
* Uncorrectable coagulopathy
* Significant active cardiac disease within the previous 6 months including: New York Heart Association (NYHA) class 4 congestive heart failure (CHF), unstable angina, or myocardial infarction
* Any condition that would prohibit the understanding or rendering of informed consent
* Any condition that in the opinion of the investigator would interfere with the participant's safety or compliance while on trial

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-11-09 (Actual); Primary Completion 2028-11 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Pathologic outcome on surveillance prostate biopsy | At year 1 and 3
  Confidence intervals for the pathologic response rate will be calculated using the Wilson score method. Pathologic response rate will be analyzed by baseline clinical and molecular characteristics using univariable and multivariable logistic regression.
Proportion of participants who go onto whole gland salvage treatment | At 3 years
  Will be estimated using the Kaplan-Meier method.
Salvage whole gland treatment free survival | At 3 years
  Will be analyzed by baseline clinical and molecular characteristics using univariable and multivariable Cox proportional hazards models.

SECONDARY OUTCOMES:
Urinary function | At 1 year
  Scores from Expanded Prostate Cancer Index Composite (EPIC-26) prostate cancer questionnaire will be used to assess urinary function.
Sexual function | At 1 year
  Scores from EPIC-26 prostate cancer questionnaire will be used to assess sexual function.
Quality of life | At 1 year
  Scores from EPIC-26 prostate cancer questionnaire will be used to assess quality of life.
Adverse events | Up to end of treatment visit, approximately 7-14 days after treatment
  Number of participants experiencing treatment-related AEs, classified by severity and grade.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Dall'Era, Principal Investigator — University of California, Davis
Locations (1):
- University of California Davis Comprehensive Cancer Center, Sacramento, California, United States